CLINICAL TRIAL: NCT02611141
Title: Retromolar Route Access With and Without A Retromolar Gap - A Visualization Study Of The Vocal Cords
Brief Title: Retromolar Route Access With and Without A Retromolar Gap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Wolfgang SCHRAMM, Ao Univ. Prof. Dr. med. univ., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1848/2015
Record Dates: First submitted 2015-11-07; First posted 2015-11-20 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Airway Management
Keywords: Retromolar Intubation

ARMS (2):
- Patient with Retromolar Gap (Other): 20 patients with a retromolar gap between the last erupted molar and the ascending ramus at the right lower mandible.
  Interventions: Procedure: Retromolar laryngoscopy and scoring of the visualisation of the vocal cords according to Cormack & Lehane
- Patient without a Retromolar Gap (Other): 20 patients without a retromolar gap between the last erupted molar and the ascending ramus at the right lower mandible.
  Interventions: Procedure: Retromolar laryngoscopy and scoring of the visualisation of the vocal cords according to Cormack & Lehane

INTERVENTIONS:
Procedure: Retromolar laryngoscopy and scoring of the visualisation of the vocal cords according to Cormack & Lehane — To facilitate the insertion of the straight blade laryngoscope (Miller #4) the head of the patient will be turned to the left side. The blade will be inserted and then pushed laterally rightwards until the retromolar space will be finally reached. Thereafter the epiglottis will be lifted up in order to achieve the best direct view to the vocal cords and scored according to Cormack & Lehane .
  This score will be assessed at least 2 minutes after muscle relaxation:
  1. Once without a backward, upward, rightwards pressure maneuver (=BURB) and immediately thereafter (i.e. 5-10 seconds later):
  2. If 100% visualization of the vocal cords is not possible a BURP maneuver will be performed and the scored again.
  Intubation will then be performed by the conventional method using a Macintosh blade #3. In the case that intubation with the conventional method is not successful the retromolar technique will be used.

SUMMARY:
Retromolar Intubation is a successful option for intubation in patients with an existing retromolar gap in the case that the conventional method fails.

Therefore the investigators want to test if the retromolar gap is essential for performing the retromolar intubation technique.

DETAILED DESCRIPTION:
For successful endotracheal intubation an optimal visualisation of the vocal cords is essential. A study comparing retromolar and conventional laryngoscopy showed in patients with an existing retromolar gap, that the retromolar technique is superior for endotracheal intubation especially in patients with a failed 'conventional' intubation attempt. The aim of the following study is to test if a retromolar gap at the right mandible is necessary for the successful performance of the retromolar laryngoscopy technique.

Therefore, 20 patients with and 20 patients without a retromolar gap will be investigated.

The anesthesiologist will visually determine the view of the vocal cords and score it according to Cormack & Lehane. For an improved view a backward, upward, right-ward pressure (BURP) will be performed, if needed, and scored again.

Finally, endotracheal intubation will be performed by the 'conventional' intubation method. If, however, intubation is not possible, then the retromolar technique will be used. In the case that both methods fail, then any (other) intubation method will (can) be used.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35kg/m2
* Elective surgery
* Absence of at least one molar of the right mandible in arm I (20 patients)

Exclusion Criteria:

* Emergency patients
* Prevalence of reflux disease
* Toothless patients
* Diaphragmatic hernia
* Patient is not sober
* Ventilation problems during induction of anaesthesia
* Patient with a tracheostomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Cormack & Lehane score (without a backward, upward, rightwards pressure maneuver) | At least 2 minutes after muscle relaxation
  After ensuring sufficient bag-mask ventilation, the scoring of the vocal cords according to Cormack & Lehane will be performed at least 2 minutes after administration of the muscle relaxant rocuronium without a backward, upward, rightwards pressure maneuver (=BURB)
Cormack & Lehane score (with a backward, upward, rightwards pressure maneuver) | Approximately 5-10 seconds after the collection of the Outcome Measure 1
  If the Outcome Measure 1 does not reveal a 100% visualization of the vocal cords, a backward, upward, rightwards pressure maneuver (BURP) maneuver will be applied and scored again according to Cormack & Lehane .
  Usually each of the two scoring procedures lasts approximately 5-10 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Ranieri D Jr, Filho SM, Batista S, do Nascimento P Jr. Comparison of Macintosh and Airtraq laryngoscopes in obese patients placed in the ramped position. Anaesthesia. 2012 Sep;67(9):980-5. doi: 10.1111/j.1365-2044.2012.07200.x. Epub 2012 Jun 1. PMID 22670846
- [Background] De Jong A, Molinari N, Conseil M, Coisel Y, Pouzeratte Y, Belafia F, Jung B, Chanques G, Jaber S. Video laryngoscopy versus direct laryngoscopy for orotracheal intubation in the intensive care unit: a systematic review and meta-analysis. Intensive Care Med. 2014 May;40(5):629-39. doi: 10.1007/s00134-014-3236-5. Epub 2014 Feb 21. PMID 24556912
- [Background] Scott J, Baker PA. How did the Macintosh laryngoscope become so popular? Paediatr Anaesth. 2009 Jul;19 Suppl 1:24-9. doi: 10.1111/j.1460-9592.2009.03026.x. PMID 19572841
- [Background] Henderson JJ. Questions about the macintosh laryngoscope and technique of laryngoscopy. Eur J Anaesthesiol. 2000 Jan;17(1):2-5. doi: 10.1046/j.1365-2346.2000.00611.x. No abstract available. PMID 10758437
- [Background] Behringer EC, Kristensen MS. Evidence for benefit vs novelty in new intubation equipment. Anaesthesia. 2011 Dec;66 Suppl 2:57-64. doi: 10.1111/j.1365-2044.2011.06935.x. PMID 22074080
- [Background] Levitan RM, Heitz JW, Sweeney M, Cooper RM. The complexities of tracheal intubation with direct laryngoscopy and alternative intubation devices. Ann Emerg Med. 2011 Mar;57(3):240-7. doi: 10.1016/j.annemergmed.2010.05.035. Epub 2010 Jul 31. PMID 20674088
- [Background] Bonfils P. [Difficult intubation in Pierre-Robin children, a new method: the retromolar route]. Anaesthesist. 1983 Jul;32(7):363-7. German. PMID 6614426
- [Background] Martinez-Lage JL, Eslava JM, Cebrecos AI, Marcos O. Retromolar intubation. J Oral Maxillofac Surg. 1998 Mar;56(3):302-5; discussion 305-6. doi: 10.1016/s0278-2391(98)90103-3. PMID 9496840